CLINICAL TRIAL: NCT02862548
Title: A Phase 2, Randomized, Open Label Study to Evaluate the Efficacy and Safety of Tenofovir Alafenamide (TAF) Versus Tenofovir Disoproxil Fumarate (TDF)-Containing Regimens in Subjects With Chronic HBV Infection and Stage 2 or Greater Chronic Kidney Disease Who Have Received a Liver Transplant
Brief Title: Efficacy and Safety of Tenofovir Alafenamide (TAF) Versus Tenofovir Disoproxil Fumarate (TDF)-Containing Regimens in Participants With Chronic Hepatitis B Virus (HBV) Infection and Stage 2 or Greater Chronic Kidney Disease Who Have Received a Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-320-3912; ACTRN12616000898459 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- TAF (Experimental): TAF 25 mg once daily for 48 weeks
  Interventions: Drug: TAF
- TDF-Containing Regimens (Active Comparator): TDF alone or in combination with other approved antivirals per local practice for 48 weeks
  Interventions: Drug: TDF; Drug: Other approved antivirals
- Optional Treatment Extension Phase (Experimental): After Week 48, participants will be eligible to receive TAF 25 mg once daily for an additional 144 weeks.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — Tablet administered orally
  Other Names: Vemlidy®
  Arms: Optional Treatment Extension Phase; TAF
Drug: TDF — Tablet administered orally
  Arms: TDF-Containing Regimens
Drug: Other approved antivirals — Other approved antivirals (such as lamivudine, entecavir, or immunoglobulin antihepatitis B) administered per local practice
  Arms: TDF-Containing Regimens

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, and efficacy of tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF)-containing regimens at Week 24 in participants with chronic hepatitis B virus (HBV) infection and Stage 2 or greater chronic kidney disease who have received a liver transplant.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures
* Documented evidence of chronic HBV infection prior to transplantation
* Primary or secondary (re-transplant), liver alone or liver and kidney transplant recipient from deceased or living donor
* Liver Transplant ≥ 12 weeks prior to screening
* Maintained on TDF alone or in combination with other approved antivirals for HBV prophylaxis or treatment
* Have been on approved HBV oral antiviral (OAV) treatment for at least 12 weeks post-transplant prior to screening, with HBV DNA < lower limit of quantification (LLOQ) at screening
* Screening estimated glomerular filtration rate using the chronic kidney disease epidemiology collaboration (eGFR_CKD-EPI) < 90 ml/min/1.73m^2
* Male participants and female participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Women considered of child bearing potential must have a negative serum pregnancy test at Screening and a negative urine test at Baseline before dosing
* Must be willing and able to comply with all study requirements

Key Exclusion Criteria:

* Multi-organ transplant that includes heart or lung recipient (participants who have their liver transplant as part of a liver-kidney dual transplant are eligible to enroll)
* Participants with history of de novo or recurrent hepatocellular carcinoma (HCC) post-transplant and at screening
* Histological evidence of unresolved transplant rejection
* Current, uncontrolled ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome, hepatopulmonary syndrome, or other signs of decompensated cirrhosis
* Participants meeting any of the following laboratory parameters at screening:

  * Alanine aminotransferase (ALT) > 10 × the upper limit of normal (ULN)
  * International normalized ratio (INR) > 1.5 × ULN unless the participant is stable on anticoagulant regimen affecting INR
  * Albumin < 3.0 g/dL
  * Direct bilirubin ≥ 4 × ULN
  * Platelet count < 50,000/mL
* Co-infection with HIV or hepatitis C virus (HCV)
* Recent (within 4 weeks of Screening) episode or infection requiring systemic antibiotics
* Use of any prohibited medications listed within 28 days of the Baseline/Day 1 visit
* Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (e.g., basal cell skin cancer, etc.) or hepatocellular carcinoma. Participants under evaluation for possible malignancy are not eligible
* Significant cardiovascular, pulmonary, or neurological disease
* Use of investigational agents within 3 months of screening, unless allowed by the Sponsor
* Use of any prohibited medications
* Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance
* Known hypersensitivity to study drugs, metabolites or formulation excipients
* Lactating females or those who may wish to become pregnant during the course of the study

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a study site in New Zealand. The first participant was screened on 16 September 2016. The last study visit occurred on 05 May 2021.
Pre-assignment Details: 57 participants were screened.
Groups:
- TAF 25 mg: Randomized Phase: Tenofovir alafenamide (TAF) 25 mg tablet orally once daily for 48 weeks
  Open-Label Extension (OLE) Phase: TAF 25 mg tablet orally once daily for additional 144 weeks
- TDF-Containing Regimens: Randomized Phase: Tenofovir disoproxil fumarate (TDF) alone or in combination with other approved antivirals per local practice for 48 weeks
  OLE Phase: TAF 25 mg tablet orally once daily for additional 144 weeks
Period: Randomized Phase (Up to Week 48)
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Started | 26 | 25
Completed | 26 | 24
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: OLE Phase (Week 49 to Week 192)
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Started | 26 | 24
Completed | 23 | 23
Not Completed | 3 | 1
Not completed — Death | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew Consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Groups:
- TAF 25 mg: Randomized Phase: TAF 25 mg tablet orally once daily for 48 weeks
  OLE Phase: TAF 25 mg tablet orally once daily for additional 144 weeks
- TDF-Containing Regimens: Randomized Phase: TDF alone or in combination with other approved antivirals per local practice for 48 weeks
  OLE Phase: TAF 25 mg tablet orally once daily for additional 144 weeks
- Total: Total of all reporting groups
Arm/Group | TAF 25 mg | TDF-Containing Regimens | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.6) | 62 (8.3) | 60 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 16 | 22 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 7 | 10 | 17
  Race: Black or African American | 1 | 0 | 1
  Race: Native Hawaiian or Pacific Islander | 15 | 12 | 27
  Race: White | 2 | 3 | 5
  Race: Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 26 | 25 | 51
HBV Deoxy Ribonucleic Acid (DNA) [Mean (Standard Deviation); unit: International unit per mL (IU/mL)] | 19.0 (0.00) | 19.0 (0.00) | 19.0 (0.00)
eGFR by CKD-EPI Creatinine [Median (Standard Deviation); unit: mL/minute/1.73 square meter(m^2)] | 52.3 (12.31) | 52.4 (12.74) | 52.4 (12.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Estimated Glomerular Filtration Rate (eGFR) at Week 24 Using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation
Time Frame: Baseline, Week 24
Population: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Groups:
- TAF 25 mg: Randomized Phase: TAF 25 mg tablet orally once daily for 48 weeks
- TDF-Containing Regimens: Randomized Phase: TDF alone or in combination with other approved antivirals per local practice for 48 weeks
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 25
mL/min/1.73 m^2 | 2.13 (6.011) | 1.87 (6.553)

2. Primary Outcome: Percentage of Participants With HBV DNA < 20 IU/mL at Week 24
Time Frame: Week 24
Population: Full Analysis Set included all randomized participants who have received at least 1 dose of study drug. The missing = failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 25
percentage of participants | 100.0 | 100.0

3. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 24
Time Frame: Baseline, Week 24
Population: Hip dual energy x-ray absorptiometry (DXA) Analysis Set included participants who were randomized and had received at least 1 dose of study drug, and had nonmissing baseline hip BMD values.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 25
percent change | 0.478 (1.6342) | 0.452 (2.1380)

4. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 23
percent change | 1.253 (1.9774) | -0.413 (2.6361)

5. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 24
Time Frame: Baseline, Week 24
Population: Spine DXA Analysis Set included participants who were randomized and had received at least 1 dose of study drug, and had nonmissing baseline spine BMD values.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 24
percent change | 0.799 (2.5563) | -0.188 (2.5890)

6. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 21
percent change | 1.454 (4.5405) | -1.082 (3.0031)

7. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 25
mg/dL | -0.043 (0.1434) | -0.040 (0.1623)

8. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 22
mg/dL | -0.052 (0.2233) | -0.058 (0.2158)

9. Secondary Outcome: Change From Baseline in Serum eGFR_CKD-EPI at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 22
mL/min/1.73 m^2 | 3.01 (9.385) | 2.09 (9.209)

10. Secondary Outcome: Percentage of Participants With HBV DNA < 20 IU/mL at Week 48
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed. The missing = failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF-Containing Regimens
Number analyzed (Participants) | 26 | 25
percentage of participants | 100.0 | 88.0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Randomization up to last follow up visit (maximum 236.7 weeks); Adverse Events: First dose date up to last dose date plus 30 days (maximum 225.9 weeks)
Description: All-Cause Mortality: Randomized Analysis Set included all participants who were randomized into the study.
  Adverse Events: Safety Analysis Set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Randomized Phase: TAF 25 mg: TAF 25 mg tablet orally once daily for 48 weeks
- Randomized Phase: TDF-Containing Regimens: TDF alone or in combination with other approved antivirals per local practice for 48 weeks
- OLE Phase: TAF 25 mg From TAF: Participants who received TAF 25 mg in randomized phase received TAF 25 mg tablet orally once daily for additional 144 weeks in OLE phase.
- OLE Phase: TAF 25 mg From TDF: Participants who received TDF alone o in combination with approved antivirals per local practice in randomized phase received TAF 25 mg tablet orally once daily for additional 144 weeks in OLE phase.
Arm/Group | Randomized Phase: TAF 25 mg | Randomized Phase: TDF-Containing Regimens | OLE Phase: TAF 25 mg From TAF | OLE Phase: TAF 25 mg From TDF
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/25 | 2/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/26 | 7/25 | 8/26 | 8/24
Other Adverse Events (participants affected / at risk) | 19/26 | 17/25 | 22/26 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: TAF 25 mg (N=26) | Randomized Phase: TDF-Containing Regimens (N=25) | OLE Phase: TAF 25 mg From TAF (N=26) | OLE Phase: TAF 25 mg From TDF (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 2 | 2 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic infarction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 0 | 1
Disseminated cryptococcosis (Infections and infestations) | 0 | 0 | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Disseminated varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 2
Osteomyelitis fungal (Infections and infestations) | 0 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Complications of transplanted liver (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 4
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: TAF 25 mg (N=26) | Randomized Phase: TDF-Containing Regimens (N=25) | OLE Phase: TAF 25 mg From TAF (N=26) | OLE Phase: TAF 25 mg From TDF (N=24)
Cataract (Eye disorders) | 0 | 2 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 1 | 0
Influenza like illness (General disorders) | 2 | 5 | 1 | 2
Pyrexia (General disorders) | 3 | 3 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Bone density decreased (Investigations) | 3 | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 2
Headache (Nervous system disorders) | 4 | 2 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 2 | 2 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (6):
  • Study Protocol: Original (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02862548/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT02862548/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT02862548/Prot_002.pdf
  • Study Protocol: Amendment 3 (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02862548/Prot_005.pdf
  • Statistical Analysis Plan: Week 24 Analysis (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT02862548/SAP_006.pdf
  • Statistical Analysis Plan: Final Analysis (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT02862548/SAP_007.pdf